CLINICAL TRIAL: NCT02237963
Title: Influence of the Surgical Approach on the Development of a Chronic Pain After Thoracic Surgery
Acronym: IncisionPain
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/50; 2013- A01641-44 (Other: ANSM)
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Posterolateral thoracotomy: Surgeons perform a posterolateral thoracotomy
  Interventions: Procedure: Posterolateral thoracotomy
- Axillary thoracotomy: Surgeons perform an axillary thoracotomy
  Interventions: Procedure: Axillary thoracotomy

INTERVENTIONS:
Procedure: Posterolateral thoracotomy
  Groups: Posterolateral thoracotomy
Procedure: Axillary thoracotomy
  Groups: Axillary thoracotomy

SUMMARY:
The prevalence of chronic pain after a thoracotomy is around 48 %. This research focuses on the surgical approach. The posterolateral approach is compared to the axillary approach especially in term of development of a chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thoracic surgery intervention by posterolateral or axillary thoracotomy, having no exclusion criteria for the study,

Exclusion Criteria:

* planned surgery by thoracoscopy or extended surgery,
* mental disability,
* vulnerable person within the meaning of French law,
* inability to communicate by phone,
* poor understanding of French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing thoracic surgery by posterolateral or axillary thoracotomy, having no exclusion criteria for the study,
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Chronic pain | 4 months
  Prevalence of pain 4 months after surgery. Pain is evaluated using a numeric scale ranging from 0 (no pain) to 10 (maximal pain)

SECONDARY OUTCOMES:
Early postoperative pain | 7 days
  Evolution of pain from postoperative day 1 to postoperative day 6 ("pain trajectory") Prevalence of pain 5 to 7 days after surgery. Pain is evaluated using a numeric scale ranging from 0 (no pain) to 10 (maximal pain).
  Clinical examination to detect modification of skin sensibility
Characteristics of chronic pain | 4 months
  Characteristics are notably:
  * its localization and intensity,
  * its neuropathic origin,
  * its impact on daily life,
  * required analgesic treatment,
  * need for a specific pain consultation
Quality of life | 4 months
  Specific questionnaire
Catastrophism | 4 months
  Score of Sullivan
Anxiety | 4 months
  Stai trait
Preventive role of epidural analgesia | 4 months
  Proportion of patients with chronic pain in each cohort who had had a postoperative thoracic epidural analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Michel-Cherqui, MD, Principal Investigator — Hôpital Foch
Locations (1):
- Hopital Foch, Suresnes, France

REFERENCES:
- [Background] Ringsted TK, Wildgaard K, Kreiner S, Kehlet H. Pain-related impairment of daily activities after thoracic surgery: a questionnaire validation. Clin J Pain. 2013 Sep;29(9):791-9. doi: 10.1097/AJP.0b013e318278d4e2. PMID 23370071